CLINICAL TRIAL: NCT04958434
Title: A Phase 1, First in Human, Open-label, Dose Escalation and Dose Expansion Study of TST005 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of TST005 in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Corporate Decision
Sponsor: Suzhou Transcenta Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TST005-1001
Record Dates: First submitted 2021-06-17; First posted 2021-07-12 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-08

CONDITIONS: Locally Advanced or Metastatic Cancers; Metastatic Human Papillomavirus-Related Malignant Neoplasm
Keywords: PD-L1, TGF-B
MeSH Terms: conditions — Neoplasms; Camurati-Engelmann Syndrome

STUDY DESIGN:
Intervention Model Description: Part A - Q3w 3+3 design dose escalation Part B - Dose expansion of approximately 30 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A - Dose Escalation (Experimental): Dosed every 3 weeks IV with TST005, starting dose is 1 mg/kg, and 5 dose levels will be tested.
  Interventions: Drug: TST005
- Part B - Dose Expansion (Experimental): Participants with any kind of advanced or HPV metastatic solid tumors dosed Q3W with the Part A Q3W recommended dose of TST005
  Interventions: Drug: TST005

INTERVENTIONS:
Drug: TST005 — TST005 is a bifunctional human immunoglobulin G1 (IgG1) monoclonal

SUMMARY:
This is an open label Phase 1, first-in-human (FIH) study of TST005, a bi-specific antibody consisting of a PD-L1 monoclonal antibody (mAb) and a transforming growth factor beta (TGF-β) trap in subjects with locally advanced or metastatic cancers

DETAILED DESCRIPTION:
The study has 2 parts. Part A is a dose escalation portion where the patients will be doses every three weeks following an accelerated 3+3 design. This portion will enroll approximately 25 patients with locally advanced or metastatic cancers.

Part B is an expansion portion where approximately 30 additional patients will be dosed at the recommended dose level every 3 weeks. This part will include patients with locally advanced or metastatic HPV related malignancies.

The trial will last approximately 2 years, with assessments including safety labs, ECGs, PKs and PDs and CT/MRI tumor assessments, based on the Q3W dosing schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide signed and dated informed consent
2. Patients with histologically or cytologically confirmed, locally advanced or metastatic solid tumors, evaluable by RECIST v1.1. (Part B includes metastatic HPV+ malignancies)
3. Subject who has tumor progression during or after prior therapy and for whom no standard therapy exists that would confer clinical benefit.
4. At least one measurable lesion per RECIST 1.1 (Part B only).
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS)0~1.
6. Provide archived tumor tissue samples
7. Adequate organ function

Exclusion Criteria:

1. Concurrent malignancy within 3 years prior to entry other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma, prostate cancer not requiring treatment (with or without resection), ductal carcinoma in situ of the breast, or ≤ T1 urothelial carcinoma.
2. Untreated or symptomatic central nervous system (CNS) metastases.
3. Any unresolved Grade 2 or greater toxicity from previous anticancer therapy except alopecia.
4. Active leptomeningeal disease.
5. Active autoimmune diseases or history of autoimmune diseases that may relapse, with the following exceptions:

   * Controlled type 1 diabetes
   * Hypothyroidism (provided it is managed with hormone-replacement therapy only)
   * Controlled celiac disease
   * Skin diseases not requiring systemic treatment (eg, vitiligo, psoriasis, or alopecia)
   * Any other disease that is not expected to recur in the absence of external triggering factors
6. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before the first dose of investigational product, with the following exceptions:

   * Adrenal replacement steroid (dose ≤ 10 mg daily of prednisone or equivalent)
   * Topical, ocular, intra-articular, intranasal, or inhalational corticosteroid with minimal systemic absorption
   * Short course (≤ 7 days) of corticosteroid prescribed prophylactically (eg, for contrast dye allergy) or for the treatment of a non-autoimmune condition (eg, delayed-type hypersensitivity reaction caused by contact allergen)
7. History of interstitial lung disease, noninfectious pneumonitis, or uncontrolled lung diseases, including but not limited to pulmonary fibrosis, active pneumonitis.
8. Severe cardiovascular disease, including cerebrovascular accident, transient ischemic attack, myocardial infarction, or unstable angina, New York Heart Association class III or IV heart failure or uncontrolled arrhythmia within 6 months of first dose.
9. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy within 2 weeks of screening.
10. Clinically significant bleeding within three months of the first dose.
11. Uncontrolled hypertension, defined as systolic ≥150 mm Hg or diastolic ≥90 mm Hg maintained over time and despite antihypertensive treatment.
12. Patients with QTcF > 480 ms on screening ECG or with a history of additional risk factors for TdP (e.g., heart failure, hypokalemia，family history of Long QT Syndrome)
13. Pregnant or nursing.
14. Known human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
15. A serious nonmalignant disease (e.g., psychiatric, substance abuse, uncontrolled intercurrent illness, etc.) that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.
16. Any other condition that, in the opinion of the Investigator, would prohibit the subject from participating in the study.
17. Active autoimmune disease requiring systemic therapy in the last 2 years prior to the first dose (i.e., with use of disease modifying agents, systemic corticosteroids or immunosuppressive drug).

    • Subjects with Type 1 diabetes mellitus (TD1M), hypothyroidism requiring only hormone replacement, or skin disorders not requiring systemic treatment are permitted to enroll.
18. A history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
19. < 4 weeks after any major procedures/surgery; clinically significant unhealed wound; any unhealed ulceration in GI prior to first dose of TST005.
20. History of severe immune-related adverse effects from checkpoint inhibitor (CPI) therapy (NCI CTCAE Grade 3 or 4) with the exception of endocrinopathy managed with replacement therapy or subjects who discontinued CPI therapy for CPI-associated toxicity or intolerability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Part A - Determine the maximum tolerated dose (MTD) or recommended Phase 2 dose(s) (RP2D) | Up to 90 days following last dose
  As measured by the number of participants experiencing a dose limiting toxicity (DLT) in each dosing cohort
Part B - Patient safety as characterized by frequency and severity of adverse events | Up to 90 days following last dose
  Characterize the safety profile of TST005 including the frequency and severity of treatment-emergent adverse events.

SECONDARY OUTCOMES:
Part A - Area under Plasma concentration vs. time curve (AUC) for TST005 | Up to 90 days following last dose
  Observe changes in AUC over time
Part A - Peak Plasma concentration (Cmax) for TST005 | Up to 90 days following last dose
  Observe the maximum serum concentration
Part A - Time to maximum observed serum (Tmax) for TST005 | Up to 90 days following last dose
  Tmax is the time in hours / days for TST005 to reach the maximum concentration after administration
Part A - Terminal half-life of TST005 | Up to 90 days following last dose
  Time for serum level to decrease by 1/2 during the terminal elimination phase
Immunogenicity of TST005 | Up to 90 days following last dose
  To determine if the formation of Anti-drug antibodies (ADA) or neutralizing antibodies (NAb) against TST005 are observed
Part B - Assess the Objective response rate (ORR) of TST005 | Up to 90 days following last dose
  as measured by RECIST v 1.1 and iRECIST
Part B - Assess the Disease Control rate (DCR) of TST005 | Up to 90 days following last dose
  Percentage of patients that exhibit stable disease (SD), + partial response (PR), + complete response (CR)
Part B - Assess the Duration of Response of TST005 | Up to 90 days following last dose
  Measured by the time a patient shows response
Part B - Assess the Time to Response (TTR) of TST005 | Up to 90 days following last dose
  Measured by the average time patients show a response to TST005
Part B - Assess the Progression -free Survival (PFS) of TST005 | Up to 90 days following last dose
  Measured by the average time before patients show signs of disease progression after receiving TST005
Part B - Assess the Overall Survival (OS) of TST005 | Up to 90 days following last dose
  Time between treatment of TST005 and death for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Qi, MD, Study Director — Suzhou Transcenta Therapeutics Co., Ltd.
Locations (3):
- United States (3):
  - Gabrail Cancer Center, Canton, Ohio
  - Mary Crowley Cancer Research, Dallas, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) will not be shared to other researchers